CLINICAL TRIAL: NCT00504504
Title: A Phase II Study of Rituximab + ABVD for Patients With Hodgkin's Disease
Brief Title: Rituximab and ABVD for Hodgkin's Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-218
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-05

CONDITIONS: Lymphoma
Keywords: Hodgkin's Disease; Lymphoma; Rituximab; Rituxan; Adriamycin; Doxorubicin; Rubex; Bleomycin; Bleomycin sulfate; Blenoxane; BLM; Dacarbazine; DTIC; DTIC-Dome; Vincristine; Vinblastine; Vinblastine Sulfate; ABVD; ABVD Chemotherapy Treatment
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Rituximab; Doxorubicin; Bleomycin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab + ABVD Chemotherapy (Experimental): Rituximab 375 mg/m^2 by vein (IV) over 3 to 8 hours weekly for 6 weeks in a row. ABVD Chemo: Adriamycin 25 mg/m^2 IV, Bleomycin 10 U/m^2 IV, Vinblastine 6 mg/m^2 IV, DTIC 375 mg/m^2 IV. Each but Rituximab over 3 hours every other week for a total of 12 treatments.
  Interventions: Drug: Rituximab; Drug: Adriamycin; Drug: Bleomycin; Drug: Vinblastine; Drug: Dacarbazine (DTIC)

INTERVENTIONS:
Drug: Rituximab — 375 mg/m^2 by vein over 3 to 8 hours weekly for 6 weeks in a row.
  Other Names: Rituxan
Drug: Adriamycin — 25 mg/m^2 injected by vein over 3 hours every other week for a total of 12 treatments.
  Other Names: Doxorubicin; Rubex
Drug: Bleomycin — 10 U/m^2 injected by vein over 3 hours every other week for a total of 12 treatments.
  Other Names: Bleomycin sulfate; Blenoxane; BLM
Drug: Vinblastine — 6 mg/m^2 injected by vein over 3 hours every other week for a total of 12 treatments.
  Other Names: Vinblastine Sulfate; Velban
Drug: Dacarbazine (DTIC) — 375 mg/m^2 injected by vein over 3 hours every other week for a total of 12 treatments.
  Other Names: DTIC-Dome

SUMMARY:
Primary Objective:

- To determine the feasibility, toxicity, and efficacy of Rituximab with standard dose ABVD combination chemotherapy.

ABVD combination chemotherapy consists of Adriamycin, Bleomycin, Vinblastine and DTIC.

DETAILED DESCRIPTION:
Before treatment starts, patients will have a physical exam. Bone marrow samples will be taken. Blood samples (4 to 8 tablespoons) will be taken before and during the study. A chest x-ray, CT scans of the abdomen and pelvis, and a gallium scan will be done if necessary.

Patients in this study will receive rituximab by vein over 3 to 8 hours weekly for 6 weeks in a row. ABVD will be injected over 3 hours every other week for a total of 12 treatments. On the cycles where both rituximab and ABVD are given, rituximab will be given on day 1, and ABVD will be given on day 2. Response to therapy will be determined after 3 months and at the end of therapy (6 months). At the end, patients may receive radiation therapy to areas of large masses. All treatments can be given in an outpatient setting.

Scans and x-rays will be repeated if needed after completion of therapy and every 3 months from then on. If tumors do not shrink after 3 months of therapy, patients will be offered a different treatment.

This is an investigational study. Although ABVD is considered the standard treatment for patients with Hodgkin's disease, the combination of ABVD with rituximab is considered investigational. All drugs involved in this study are commercially available and are approved by the FDA. Up to 85 patients will take part in this study. All will be enrolled at M. D. Anderson. This protocol is partially funded by a research grant from Genentech.

ELIGIBILITY:
Inclusion Criteria:

1. Hodgkin's disease patients who relapse after radiation therapy alone and previously untreated patients with stage II bulky, III and IV who are eligible for ABVD.
2. Must have histologically proven diagnosis of Hodgkin's disease (Nodular sclerosis or mixed cellularity).
3. Must have bidimensionally measurable disease.
4. Must sign a consent form.
5. Must be older than 16 years of age.
6. Must have adequate bone marrow reserve (ANC > 1,000/microL, Platelet > 100,000/microL
7. Left Ventricular Ejection Fraction (LVEF) >/= 50% by multigated acquisition (MUGA) scan or echocardiogram.
8. Serum creatinine < 2 mg/dl, serum bilirubin < 2 mg/dl

Exclusion Criteria:

1. HIV positive.
2. Pregnant women and women of child bearing age who are not practicing adequate contraception.
3. Prior chemotherapy.
4. Severe pulmonary disease including Chronic obstructive pulmonary disease (COPD) and asthma.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2001-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD . Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Younes A, Oki Y, McLaughlin P, Copeland AR, Goy A, Pro B, Feng L, Yuan Y, Chuang HH, Macapinlac HA, Hagemeister F, Romaguera J, Samaniego F, Fanale MA, Dabaja BS, Rodriguez MA, Dang N, Kwak LW, Neelapu SS, Fayad LE. Phase 2 study of rituximab plus ABVD in patients with newly diagnosed classical Hodgkin lymphoma. Blood. 2012 May 3;119(18):4123-8. doi: 10.1182/blood-2012-01-405456. Epub 2012 Feb 27. PMID 22371887
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 09, 2001 to August 29, 2007. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 85 participants enrolled, three participants were excluded prior to assignment to groups as ineligible.
Period: Overall Study
Arm/Group | Rituximab + ABVD Chemotherapy
Started | 82
Completed | 82
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab + ABVD Chemotherapy
Number analyzed (Participants) | 82
Age Continuous [Median (Full Range); unit: years] | 32 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 82

OUTCOME MEASURES:

1. Primary Outcome: 5-year Failure-free Survival Rate for Participants With Hodgkin's Disease Given Rituximab With ABVD
Description: Five year Event Free Survival (EFS) is proportion of surviving participants who remain event free out of total participants at 5 years after receiving Rituximab + ABVD (RABVD). Event-free Survival (EFS) analyzed every 6 months.
Time Frame: Baseline to 5 Years or until disease progression
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + ABVD Chemotherapy
Number analyzed (Participants) | 82
percentage of participants | 83

ADVERSE EVENTS:
Time Frame: 6 years and 5 months
Arm/Group | Rituximab + ABVD Chemotherapy
Serious Adverse Events (participants affected / at risk) | 40/82
Other Adverse Events (participants affected / at risk) | 82/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + ABVD Chemotherapy (N=82)
Fatigue (General disorders) | 7
Pain (General disorders) | 5
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Neuropathy (Nervous system disorders) | 1
Granuloctopenia (Blood and lymphatic system disorders) | 18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + ABVD Chemotherapy (N=82)
Fatigue (General disorders) | 32
Pain (General disorders) | 28
Alopecia (General disorders) | 35
Nausea (Gastrointestinal disorders) | 45
Vomiting (Gastrointestinal disorders) | 28
Diarrhea (Gastrointestinal disorders) | 16
Constipation (Gastrointestinal disorders) | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Neuropathy (Nervous system disorders) | 25
Granuloctopenia (Blood and lymphatic system disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No